CLINICAL TRIAL: NCT03799874
Title: A Phase II Trial of Inhaled Carbon Monoxide for the Treatment of Acute Respiratory Distress Syndrome (ARDS)
Brief Title: Safety and Efficacy Study of Inhaled Carbon Monoxide to Treat Acute Respiratory Distress Syndrome (ARDS)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Massachusetts General Hospital (Other); Weill Medical College of Cornell University (Other); Duke University (Other); Durham VA Medical Center (U.S. Federal Agency); New York Presbyterian Brooklyn Methodist Hospital (Other); Duke Regional Hospital (Other); U.S. Army Medical Research Acquisition Activity (U.S. Federal Agency); Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Rebecca Baron, Associate Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018P002051; CDMRP-PR171025, W81XWH1810667 (Other Grant/Funding Number: United States Army Medical Research Acquisition Activity)
Record Dates: First submitted 2018-12-06; First posted 2019-01-10 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: The study drug will be blinded to the study staff using identical tanks containing either CO or placebo air. The administering respiratory therapist (RT) and a physician study staff member will be unblinded to the treatment assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Inhaled Carbon Monoxide (Experimental): Inhaled Carbon Monoxide at 200 ppm for up to 90 minutes daily for 3 days.
  Interventions: Drug: Inhaled Carbon Monoxide at 200 ppm
- Medical air (Placebo Comparator): Inhaled Medical Air for up to 90 minutes daily for 3 days.
  Interventions: Other: Inhaled Medical air

INTERVENTIONS:
Drug: Inhaled Carbon Monoxide at 200 ppm — Inhaled Carbon Monoxide at 200 ppm for 90 minutes daily for 3 days.
  Other Names: iCO
  Arms: Inhaled Carbon Monoxide
Other: Inhaled Medical air — Inhaled Medical Air for up to 90 minutes daily for 3 days.
  Arms: Medical air

SUMMARY:
This study will be a multi-center, prospective, randomized, partially double-blind, placebo-controlled Phase II clinical trial of inhaled CO (iCO) for the treatment of ARDS. The trial will be conducted at 7 tertiary care medical centers including Weill Cornell Medicine/NewYork-Presbyterian Hospital, Brigham and Women's Hospital (BWH), Massachusetts General Hospital (MGH), Duke University Hospital, Durham Veterans Administration Medical Center, New York-Presbyterian Brooklyn Methodist Hospital, and Duke Regional Hospital. The purpose of this study is to evaluate the safety, tolerability, and efficacy of inhaled carbon monoxide (iCO) for the treatment of ARDS and to examine the biologic readouts of low dose iCO therapy in patients with ARDS

DETAILED DESCRIPTION:
Acute respiratory distress syndrome (ARDS) is a devastating disease affecting military, veteran, and civilian populations. ARDS is a syndrome of severe acute lung inflammation and hypoxemic respiratory failure with an incidence of 180,000 cases annually in the United States. Despite recent advances in critical care management and lung protective ventilation strategies, ARDS morbidity and mortality remain unacceptably high. The lack of specific effective therapies for ARDS indicates a need for new treatments that target novel pathways. Carbon monoxide (CO) represents a novel therapeutic modality in ARDS based on data obtained in experimental models of ARDS over the past decade.

CO has been shown to be protective in experimental models of acute lung injury (ALI) and sepsis. Furthermore, multiple human studies have demonstrated that experimental administration of several different concentrations of CO is well tolerated and that low dose inhaled CO can be safely administered to subjects in a controlled research environment. The investigators have previously conducted a Phase I trial of low dose iCO in ARDS which demonstrated that precise administration of low dose iCO (100 and 200 ppm) is feasible, well-tolerated, and safe in patients with sepsis-induced ARDS.

The purpose of this study is to assess the safety and efficacy of low dose inhaled carbon monoxide (iCO) therapy in mechanically ventilated patients with ARDS.

ELIGIBILITY:
Inclusion Criteria:

All intubated patients ≥ 18 years old with ARDS

1. ARDS is defined when all four of the following criteria are met:

   1. A PaO2/FiO2 ratio ≤ 300 with at least 5 cm H2O positive end-expiratory airway pressure (PEEP)
   2. Bilateral opacities on frontal chest radiograph (not fully explained by effusions, lobar/lung collapse, or nodules) within 1 week of a known clinical insult or new or worsening respiratory symptoms
   3. A need for positive pressure ventilation by an endotracheal or tracheal tube
   4. Respiratory failure not fully explained by cardiac failure or fluid overload; need objective assessment (e.g., echocardiography) to exclude hydrostatic edema if no risk factor present.
2. ARDS onset is defined as the time the last of criteria 1-4 are met. ARDS must persist through the enrollment time window of 168 hours.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Age less than 18 years
2. Greater than 168 hours since ARDS onset
3. Pregnant or breastfeeding
4. Prisoner
5. Patient, surrogate, or physician not committed to full support (exception: a patient will not be excluded if he/she would receive all supportive care except for attempts at resuscitation from cardiac arrest)
6. No consent/inability to obtain consent or appropriate legal representative not available
7. Physician refusal to allow enrollment in the trial
8. Moribund patient not expected to survive 24 hours
9. No arterial or central line/no intent to place an arterial or central line
10. No intent/unwillingness to follow lung protective ventilation strategy
11. Severe hypoxemia defined as SpO2 < 95 or PaO2 < 90 on FiO2 ≥ 0.9
12. Hemoglobin < 7.0 g/dL
13. Subjects who are Jehovah's Witnesses or are otherwise unable or unwilling to receive blood transfusions during hospitalization
14. Acute myocardial infarction (MI) or acute coronary syndrome (ACS) within the last 90 days
15. Coronary artery bypass graft (CABG) surgery within 30 days
16. Angina pectoris or use of nitrates with activities of daily living
17. Cardiopulmonary disease classified as NYHA class IV
18. Stroke (ischemic or hemorrhagic) within the prior 1 month, cardiac arrest requiring CPR within the prior 72 hours, or inability to assess mental status following cardiac arrest
19. Burns > 40% total body surface area (TBSA)
20. Severe airway inhalational injury
21. Use of high frequency oscillatory ventilation
22. Use of extracorporeal membrane oxygenation (ECMO)
23. Concomitant use of inhaled pulmonary vasodilator therapy (eg. nitric oxide [NO] or prostaglandins)
24. Diffuse alveolar hemorrhage from vasculitis
25. Concurrent participation in other investigational drug study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Outcome: Number of pre-specified administration-related adverse events. | 7 days
  Safety of inhaled CO, defined by the incidence of pre-specified administration-related AEs (as defined below) and spontaneously reported AEs through study day 7.
  1. Acute MI within 48 hours of study drug administration
  2. Acute cerebrovascular accident (CVA) within 48 hours of study drug administration
  3. New onset atrial or ventricular arrhythmia requiring DC cardioversion within 48 hours of study drug administration
  4. Increased oxygenation requirements defined as: an increase in FiO2 of ≥ 0.2 AND increase in PEEP ≥ 5 cm H2O within 6 hours of study drug administration
  5. Increase in COHb ≥ 10%
  6. Increase in lactate by ≥ 2 mmol/L within 6 hours of study drug administration
Primary Efficacy Outcome: Change in Mitochondrial DNA (mtDNA) level from day 1 to day 5 | 5 days
  Mitochondrial DNA (mtDNA) plasma levels will be measured by quantitative PCR of human NADH dehydrogenase 1.

SECONDARY OUTCOMES:
Lung injury score (LIS) on days 1-5, and on day 7 | 7 days
  The Lung Injury Score (LIS) is a composite 4-point scoring system including the PaO2/FiO2, PEEP, quasi-static respiratory compliance, and the extent of infiltrates on the chest X-ray. Each of the four components is categorized from 0 to 4, where a higher number is worse. The total Lung Injury Score is obtained by dividing the aggregate sum by the number of components used. Previous randomized clinical trials in ARDS have shown that a decreased LIS correlates with improvement in lung physiology as well as important clinical outcomes including mortality and ventilator-free days (VFDs).
PaO2/FiO2 ratio on days 1-5, and on day 7 | 7 days
  PaO2/FiO2 will be measured daily on days 1-5 and on day 7 in ventilated subjects.
Oxygenation Index (OI) on days 1-5, and day 7 | 7 days
  The oxygenation index will be measured daily on days 1-5 and on day 7 in ventilated subjects. Oxygenation index is calculated as (FiO2 X mean airway pressure)/PaO2.
Dead Space Fraction (Vd/Vt) on days 1-3, and day 7 | 7 days
  The dead space fraction will be measured daily on days 1-3 and on day 7 in ventilated subjects.
Sequential Organ Failure Assessment (SOFA) score on days 1-5, 7, 14, 28 | 28 days
  Organ failure will be assessed using the SOFA score. SOFA scores will be assessed daily on days 1-5, and thereafter on days 7, 14, and 28, as the SOFA score has been shown to be a reliable prognostic indicator of outcomes in critically ill patients. To calculate the Sequential Organ Failure Assessment (SOFA) score, each of the six components (Respiratory, Coagulation, Liver, Cardiovascular, Central Nervous System, Renal) is categorized from 0-4, where a higher number is worse. The SOFA score (0-24) will be calculated by summing all six components.
Change in biomarkers of autophagy | 5 days
  Autophagy markers (eg. LC3B) will be measured in plasma daily on days 1-3 and on day 5.
Change in biomarkers of inflammation and inflammasome activation | 5 days
  Cytokine plasma levels (eg. IL-18) will be measured by ELISA daily on days 1-3 and on day 5.
Change in lipid mediators | 5 days
  Lipid mediators (LM) and specialized pro-resolving mediators (SPMs) will be measured in plasma using liquid chromatography-tandem mass spectrometry (LC-MS-MS) based methods daily on days 1-3 and on day 5.
Change in biomarkers of mitochondrial quality control | 5 days
  Mitochondrial quality control biomarkers (eg. Pink1, Wipi1) will be measured in peripheral blood mononuclear cells (PBMCs) daily on days 1-3 and on day 5.

OTHER OUTCOMES:
Ventilator-free days at day 28 | 28 days
  Ventilator-free days to day 28 are defined as the number of days from the time of initiating unassisted breathing to day 28 after randomization, assuming survival for at least two consecutive calendar days after initiating unassisted breathing and continued unassisted breathing to day 28. If a subject returns to assisted breathing and subsequently achieves unassisted breathing to day 28, VFDs will be counted from the end of the last period of assisted breathing to day 28. Participants who do not survive to day 28 are assigned zero ventilator-free days.
ICU-free days at day 28 | 28 days
  ICU-free days will be assessed on day 28. ICU-free days is defined as the number of days between randomization and day 28 in which the patient is in the ICU (for any part of a day).
Hospital-free days at day 60 | 60 days
  Hospital-free days will be assessed on day 60. Hospital-free days are days alive post hospital discharge through day 60. Patients who die on or prior to day 60 are assigned zero hospital-free days.
Hospital mortality to day 28 and 60 | 60 days
  Mortality will be assessed on day 28 and day 60
Montreal Cognitive Assessment- MoCA-Blind | 6 months
  The MoCA-Blind will be administered at 6 months via telephone interview to assess 4 items examining attention, verbal learning and memory, executive functions/language, and orientation. The test is scored out of 22 with 18 and above considered normal.
Hayling Sentence Completion Test | 6 months
  The Hayling Sentence Completion Test will be administered at 6 months via telephone interview. The Hayling Sentence Completion Test is a neuropsychological test consisting of two types of sentence completion. The first section is scored based on time taken to complete the sentence. The second section is scored based on time taken to complete a sentence as well as the quality of answer. These scores are combined and scaled according to age.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Baron, MD, Principal Investigator — Brigham and Women's Hospital
Locations (7):
- United States (7):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - New York-Presbyterian Brooklyn Methodist Hospital, Brooklyn, New York
  - Weill Cornell Medical College, New York, New York
  - Duke Regional Hospital, Durham, North Carolina
  - Duke University Hospital, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nakahira K, Kyung SY, Rogers AJ, Gazourian L, Youn S, Massaro AF, Quintana C, Osorio JC, Wang Z, Zhao Y, Lawler LA, Christie JD, Meyer NJ, Mc Causland FR, Waikar SS, Waxman AB, Chung RT, Bueno R, Rosas IO, Fredenburgh LE, Baron RM, Christiani DC, Hunninghake GM, Choi AM. Circulating mitochondrial DNA in patients in the ICU as a marker of mortality: derivation and validation. PLoS Med. 2013 Dec;10(12):e1001577; discussion e1001577. doi: 10.1371/journal.pmed.1001577. Epub 2013 Dec 31. PMID 24391478
- [Background] Brealey D, Brand M, Hargreaves I, Heales S, Land J, Smolenski R, Davies NA, Cooper CE, Singer M. Association between mitochondrial dysfunction and severity and outcome of septic shock. Lancet. 2002 Jul 20;360(9328):219-23. doi: 10.1016/S0140-6736(02)09459-X. PMID 12133657
- [Background] Jung SS, Moon JS, Xu JF, Ifedigbo E, Ryter SW, Choi AM, Nakahira K. Carbon monoxide negatively regulates NLRP3 inflammasome activation in macrophages. Am J Physiol Lung Cell Mol Physiol. 2015 May 15;308(10):L1058-67. doi: 10.1152/ajplung.00400.2014. Epub 2015 Mar 13. PMID 25770182
- [Background] Rhodes MA, Carraway MS, Piantadosi CA, Reynolds CM, Cherry AD, Wester TE, Natoli MJ, Massey EW, Moon RE, Suliman HB. Carbon monoxide, skeletal muscle oxidative stress, and mitochondrial biogenesis in humans. Am J Physiol Heart Circ Physiol. 2009 Jul;297(1):H392-9. doi: 10.1152/ajpheart.00164.2009. Epub 2009 May 22. PMID 19465554
- [Background] Fredenburgh LE, Kraft BD, Hess DR, Harris RS, Wolf MA, Suliman HB, Roggli VL, Davies JD, Winkler T, Stenzler A, Baron RM, Thompson BT, Choi AM, Welty-Wolf KE, Piantadosi CA. Effects of inhaled CO administration on acute lung injury in baboons with pneumococcal pneumonia. Am J Physiol Lung Cell Mol Physiol. 2015 Oct 15;309(8):L834-46. doi: 10.1152/ajplung.00240.2015. Epub 2015 Aug 28. PMID 26320156
- [Background] Hausberg M, Somers VK. Neural circulatory responses to carbon monoxide in healthy humans. Hypertension. 1997 May;29(5):1114-8. doi: 10.1161/01.hyp.29.5.1114. PMID 9149675
- [Background] Mayr FB, Spiel A, Leitner J, Marsik C, Germann P, Ullrich R, Wagner O, Jilma B. Effects of carbon monoxide inhalation during experimental endotoxemia in humans. Am J Respir Crit Care Med. 2005 Feb 15;171(4):354-60. doi: 10.1164/rccm.200404-446OC. Epub 2004 Nov 19. PMID 15557136
- [Background] Peterson JE, Stewart RD. Predicting the carboxyhemoglobin levels resulting from carbon monoxide exposures. J Appl Physiol. 1975 Oct;39(4):633-8. doi: 10.1152/jappl.1975.39.4.633. PMID 1194155
- [Background] Stewart RD, Peterson JE, Baretta ED, Bachand RT, Hosko MJ, Herrmann AA. Experimental human exposure to carbon monoxide. Arch Environ Health. 1970 Aug;21(2):154-64. doi: 10.1080/00039896.1970.10667214. No abstract available. PMID 5430001
- [Background] Zevin S, Saunders S, Gourlay SG, Jacob P, Benowitz NL. Cardiovascular effects of carbon monoxide and cigarette smoking. J Am Coll Cardiol. 2001 Nov 15;38(6):1633-8. doi: 10.1016/s0735-1097(01)01616-3. PMID 11704374
- [Background] Ren X, Dorrington KL, Robbins PA. Respiratory control in humans after 8 h of lowered arterial PO2, hemodilution, or carboxyhemoglobinemia. J Appl Physiol (1985). 2001 Apr;90(4):1189-95. doi: 10.1152/jappl.2001.90.4.1189. PMID 11247913
- [Background] Pecorella SR, Potter JV, Cherry AD, Peacher DF, Welty-Wolf KE, Moon RE, Piantadosi CA, Suliman HB. The HO-1/CO system regulates mitochondrial-capillary density relationships in human skeletal muscle. Am J Physiol Lung Cell Mol Physiol. 2015 Oct 15;309(8):L857-71. doi: 10.1152/ajplung.00104.2015. Epub 2015 Jul 17. PMID 26186946
- [Background] Fredenburgh LE, Perrella MA, Barragan-Bradford D, Hess DR, Peters E, Welty-Wolf KE, Kraft BD, Harris RS, Maurer R, Nakahira K, Oromendia C, Davies JD, Higuera A, Schiffer KT, Englert JA, Dieffenbach PB, Berlin DA, Lagambina S, Bouthot M, Sullivan AI, Nuccio PF, Kone MT, Malik MJ, Porras MAP, Finkelsztein E, Winkler T, Hurwitz S, Serhan CN, Piantadosi CA, Baron RM, Thompson BT, Choi AM. A phase I trial of low-dose inhaled carbon monoxide in sepsis-induced ARDS. JCI Insight. 2018 Dec 6;3(23):e124039. doi: 10.1172/jci.insight.124039. PMID 30518685
- [Background] Rosas IO, Goldberg HJ, Collard HR, El-Chemaly S, Flaherty K, Hunninghake GM, Lasky JA, Lederer DJ, Machado R, Martinez FJ, Maurer R, Teller D, Noth I, Peters E, Raghu G, Garcia JGN, Choi AMK. A Phase II Clinical Trial of Low-Dose Inhaled Carbon Monoxide in Idiopathic Pulmonary Fibrosis. Chest. 2018 Jan;153(1):94-104. doi: 10.1016/j.chest.2017.09.052. Epub 2017 Oct 31. PMID 29100885